CLINICAL TRIAL: NCT03690154
Title: A Phase 1, Multi-center, Open-label, Single-arm, Dose-escalation, Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of FN-1501 Monotherapy in Patients With Advanced Solid Tumors or Relapsed/Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Phase 1 Study to Evaluate FN-1501 Monotherapy in Patients With Advanced Solid Tumors and R/R AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Despite demonstrated safety and tolerability the trial was terminated early due to program re-prioritization in light of the competitive landscape.
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FN-1501-UP1
Record Dates: First submitted 2018-09-21; First posted 2018-10-01 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2022-07

CONDITIONS: Advanced Cancer; Solid Tumors; Acute Myeloid Leukemia Refractory; Acute Myeloid Leukemia, in Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FN-1501 (Experimental)
  Interventions: Drug: FN-1501

INTERVENTIONS:
Drug: FN-1501 — Eligible patients will receive a single intravenous infusion of study drug on Days 1, 3, 5, 8, 10, and 12 of a 21-day cycle. Dosing will begin at 2.5 mg once per day on the assigned days. Dose escalation will use the traditional 3+3 design and follow a modified Fibonacci sequence until MTD is reached. Increments of 33% in the dose of FN-1501 will be undertaken after reaching 30 mg/day. At least 3 patients will be enrolled in each cohort. Administration of FN-1501 will be continued until disease progression, intolerable toxicity, withdrawal of consent, or termination according to the Principal Investigator's judgment or at the sponsor's request.

SUMMARY:
This research study is being done in people with advanced-stage solid tumor cancer. Advanced stage solid tumor cancer is a cancer that forms an abnormal mass of tissue that usually does not contain cysts or liquid areas. Different types of solid tumors are named for the type of cells that form them. Examples of solid tumors include lung cancer, breast cancer, prostate cancer, kidney cancer, colorectal cancer, melanoma and sarcoma.

The purpose of this research study is to evaluate the safety of the investigational study drug, FN-1501, at different dose levels. FN-1501 has not previously been given to human subjects. It is intended for the treatment in this study of patients with advanced solid tumor cancers. This study will determine the effects, good and/or bad, on patients' cancer. The main objective of this study is to define the recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of FN-1501. The MTD is the highest dose a person can take without having bad side effects, and the RP2D will be the dose of FN-1501 used in future studies.

DETAILED DESCRIPTION:
This is a phase 1, first-in-human, open-label, multicenter, dose escalation study.

Dose escalation will follow the traditional 3+3 design. Patients will be screened for eligibility for up to 28 days prior to entry into the study. The starting dose will be 2.5 mg/day (once daily). The period for DLT assessment is 21 days from the first dose of FN-1501. Evaluation of a cohort of at least three (3) patients completing DLT assessment at any given dose level is required prior to determining the next dose level and dose regimen for the subsequent cohort.

After the first patient in the cohort receives the Cycle 1, Day 1 dose, subsequent patients in that cohort will not be dosed until the first patient has been evaluated for at least 48 hours to exclude unexpected acute toxicity. The continuous safety evaluation will be performed by investigators, the medical monitor, and the sponsor. A Safety Monitoring Committee (SMC) will determine dose levels to be administered and dose regimen during dose escalation based on the data available from the previous dose levels. If an MTD is not identified due to paucity of DLTs, the RP2D will be determined based on pharmacokinetics, safety, tolerability, and preliminary efficacy.

If a patient wishes to continuously receive study treatment on completion of Cycle 1, the patient can continue study treatment in 21-day Cycle 2 and subsequent cycles (same as Cycle 2, all of 21 days' duration), defined as administration of 3 times per week for 2 weeks followed by one week off, at the discretion of the investigator.

The primary endpoint of this study is to determine the recommended phase 2 dose (RP2D) of FN-1501 based on pharmacokinetics, safety and tolerability, as well as preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 18 years old and above
* Able to understand and sign informed consent form
* Patients with histologically or cytologically confirmed advanced solid tumors who have relapsed or refractory disease or relapsed/refractory AML for which no standard therapies expected to produce clinical benefit to the patient are available
* Patients with diagnosed solid tumors must have at least one lesion that is measurable per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
* Patients with relapsed or refractory AML must be diagnosed with AML based on World Health Organization (WHO) criteria (≥ 20% blasts in bone marrow). Patients with acute promyelocytic leukemia are excluded
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Have discontinued all previous cancer therapies for at least 21 days or 5 half-lives prior to study treatment, whichever is shorter, and recovered from the acute adverse effects of therapy
* Expected to survive at least 2 to 3 months
* LVEF ≥ 50% and QTc interval < 450 ms
* Women shall meet either of the following conditions before enrollment
* Infertile, defined as having a bilateral oophorectomy (ovariectomy), or a bilateral tubal ligation, or being post-menopausal for at least 1 year.
* For those of childbearing potential, they should have a negative serum pregnancy test during screening, agree to refrain from lactation, and use effective contraception such as hormonal methods associated with inhibition of ovulation, condom, intra-uterine device, surgical sterilization (including partner's vasectomy) or sexual abstinence during the study and 30 days after the last administration of study drug.
* Men who are engaging or plan to engage in sexual activity with a female of childbearing potential must either have a prior vasectomy or agree to use effective contraception such as condoms, sexual abstinence and appropriate methods taken by their partner(s) during the study and 90 days after the last dose.
* Patients must have adequate organ functions as indicated by the following screening laboratory values:
* Serum total bilirubin ≤ 1.5 × upper limit normal (ULN) (Serum total bilirubin can be ≤ 3.0 × ULN if patients have hemolysis or congenital hemolytic diseases)
* Creatinine < 1.5 × ULN or estimated creatinine clearance ≥ 50 mL/min
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN or

  * 5 X ULN for patient with liver metastases
* Absolute neutrophil count (ANC) ≥ 1.5×10^9/L
* Platelets ≥ 100×10^9/L
* Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L (Note: Criteria must be met without a transfusion within 2 weeks of obtaining the sample) Note: Laboratory requirements for complete blood counts (hemoglobin, ANC, and platelets) do not apply to AML patients

Exclusion Criteria:

* Participation in another therapeutic clinical trial within 3 weeks of enrollment
* A previous toxicity-related reaction towards cancer therapy have not recovered within 2 weeks of enrollment (>Grade 2 National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03)
* Having received a major surgical operation within 4 weeks of enrollment or not yet completely recovered from a previous operation
* Any serious or uncontrollable systemic disease, including but not limited to: Hypertension (after treatment, systolic blood pressure (SBP) > 180 mmHg and/or diastolic blood pressure (DBP) > 100 mmHg) and active hemorrhagic disorders; patients who are determined by investigators as otherwise not suitable for participation in this study.Note: Patients that in the judgment of the investigator have clinical signs of disease progression during the screening period (i.e.: febrile neutropenia, ascites requiring drainage, hospitalization due to worsening underlying disease, etc.) will not be eligible for participation.
* Active known infection, including hepatitis B, hepatitis C, and human immunodeficiency virus
* Primary central nervous system (CNS) tumor or CNS metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (patients with a history of CNS metastases or cord compression are allowable if they have been definitively treated and have been clinically stable for at least 3 months, and off steroids or anticonvulsants ≥ 2 weeks before first dose of study drug)
* Serious kidney injury, requiring dialysis
* Serious liver injury, and advanced liver diseases of Child-Pugh class B and C
* On medications that are strong cytochrome P450(CYP)3A inhibitors or inducers unless patients are willing and able to change to use of an equivalent medication that is not a strong CYP3A inhibitor or inducer
* Cardiac function and disease history which meets one or more of the following conditions:
* Any risk which may increase QTc interval prolongation, such as hypokalemia, hereditary long QT syndrome and taking drugs that can prolong QT interval
* Acute myocardial infarction ≤ 6 months prior to Day 1
* Clinically significant arrhythmia ≤ 6 months prior to Day 1
* Congestive heart failure ≥ Grade 3 by New York Heart Association (NYHA) ≤ 6 months prior to Day 1
* Cerebral vascular accident (CVA) ≤ 6 months prior to Day 1
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03 | From first dose until 30 days after the last dose.
To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) | During the first year.
  The recommended phase 2 dose (RP2D) of FN-1501 will be determined based on pharmacokinetics, safety and tolerability, as well as preliminary efficacy.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero to the last measurable concentration (AUC0-last) | During the first year.
Area under concentration-time curve from 0 to 24 hours (AUC(0-24)) | During the first year.
Area under the plasma concentration time curve from zero to infinity (AUC0-∞) | During the first year.
Maximum observed plasma concentration (Cmax) | During the first year.
Time to maximum observed plasma concentration (tmax) | During the first year.
Terminal half-life (t1/2) | During the first year.
Clearance (CL) | During the first year.
Apparent volume of distribution (Vd) | During the first year.
Measurement of anti-tumor activity of FN-1501 according to RECIST version 1.1 (solid tumor) | During the first year.
Measurement of anti-tumor activity of FN-1501 including but not limited to CT/MRI images | During the first year.

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Min Hui, MD, PhD, Study Director — Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd.
Locations (3):
- United States (2):
  - KUMC Cancer Center, Fairway, Kansas
  - Karmanos Cancer Institute, Detroit, Michigan
- Cabrini Malvern Hospital, Malvern, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT03690154/Prot_001.pdf